CLINICAL TRIAL: NCT05731700
Title: Everolimus-Coated Percutaneous Transluminal Coronary Angioplasty Catheter First in Human Clinical Investigation: A Clinical Evaluation in the Treatment of Subjects With In-Stent Restenosis of Previously-treated Coronary Artery Lesions
Brief Title: CVT-ISR First in Human Trial for Coronary In-Stent Restenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP1125
Record Dates: First submitted 2023-01-25; First posted 2023-02-16 (Actual); Results first posted 2025-05-15 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: In-stent Restenosis
Keywords: TP1125; Coronary; CVT; CVT-ISR

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Drug eluting balloon (Experimental): Treatment of a single in-stent restenosis coronary artery lesion with drug eluting balloon
  Interventions: Device: Drug Eluting Balloon

INTERVENTIONS:
Device: Drug Eluting Balloon — PCI of in-stent restenosis

SUMMARY:
The goal of this first in human study is to assess the safety and inhibition of restenosis of the CVT Everolimus-coated PTCA Catheter in the treatment of subjects presenting in-stent restenotic lesions in native coronary arteries.

DETAILED DESCRIPTION:
The CVT-ISR Trial is a prospective, multi-center, open, single arm study enrolling subjects with visually estimated nominal vessel diameter ≥2.0 mm and ≤3.5mm and lesion length ≤24 mm receiving up to two (2) CVT Everolimus CVT EVE-PTCA Catheters.

An angiographic follow up, in combination with either Intravascular Ultrasound (IVUS) or Optical Coherence Tomography (OCT), follow-up, will be carried out in a subset of 25 patients at 180 days following the index procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be at least 18 years of age.
2. Subject or his/her legally authorized representative provides written informed consent prior to any clinical investigation related procedure, as approved by the appropriate Ethics Committee of the respective clinical site.
3. Subject must agree to undergo all clinical investigation plan-required follow-up visits, angiograms, IVUS/OCT and examinations.

Angiographic Inclusion Criteria

1. Target lesion must be located within a stent (bare metal or drug eluting) placed in a native epicardial coronary vessel with visually estimated nominal vessel diameter of ≥2.0mm and ≤3.5mm.
2. Target lesion must measure ≤24 mm in length by visual estimation.
3. The target lesion must be with a visually estimated stenosis of ≥50% and < 100% with a TIMI flow of ≥1.
4. Non-clinical investigation, percutaneous intervention for lesions in a non-target vessel is allowed if done ≥90 days prior to or planned to be done 6 months after the index procedure.
5. Non-clinical investigation, percutaneous intervention for lesions in the target vessel is allowed if planned to be done 6 months after the index procedure.

Exclusion Criteria:

1. Subject with known diagnosis of acute myocardial infarction (AMI) within 30 days preceding the index procedure and CK-MB or troponin have not returned within normal limits at the time of procedure.
2. The subject is currently experiencing clinical symptoms consistent with AMI.
3. Subject has current unstable arrhythmia.
4. Subject has a known left ventricular ejection fraction (LVEF) <25%.
5. Subject has a known hypersensitivity or contraindication to aspirin, both heparin and bivalirudin, both clopidogrel and ticlopidine and structurally related compounds, everolimus, or contrast sensitivity that cannot be adequately pre-medicated.
6. Subject has known renal insufficiency (e.g., serum creatinine > 2.5 mg/dL, (i.e. 221 µmol/L) within 7 days prior to index procedure or creatinine clearance <30mL/min or subject is on dialysis.
7. Subject has a history of bleeding diathesis or coagulopathy or will refuse blood transfusions.
8. Subject has had a cerebrovascular accident (CVA) or transient ischemic neurological attack (TIA) within the past six months.
9. Subject has other medical illness (e.g., cancer or congestive heart failure) or known history of substance abuse (alcohol, cocaine, heroin etc.) that may cause non-compliance with the clinical investigation plan, confound the data interpretation or is associated with a limited life expectancy (i.e., less than one year).
10. Subject is already participating in another clinical investigation that has not yet reached its primary endpoint.
11. Subject is not, in the opinion of the investigator, an acceptable candidate to participate in the study.
12. In-stent lesions for stent are located within an arterial or saphenous vein graft or stent used to treat a previous ISR.
13. The target vessel contains visible thrombus.
14. Pregnant or lactating females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2022-09-19 (Actual); Study Completion 2025-05-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- France (3):
  - Groupe Hospitalier Mutualiste de Grenoble, Grenoble
  - L'Hôpital Privé du Confluent, Nantes
  - Clinique Pasteur, Toulouse
- Georgia (2):
  - Tbilisi Heart and Vascular Clinic, Tbilisi
  - Georgian Israeli Research Medical Centre Helsicore, Tbilisi
- Vilniaus universiteto ligoninė Santaros klinikos, Vilnius, Lithuania
- Spain (3):
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario La Paz, Madrid

REFERENCES:
- [Derived] Alfonso F, Shaburishvili T, Farah B, Gogorishvili I, Monsegu J, Baranauskas A, Bressollette E, Shaburishvili G, Cuesta J, Rivero F, Moreno R, Sabate M. First-in-man study of a novel everolimus-coated balloon for the treatment of coronary in-stent restenosis. Coron Artery Dis. 2025 Mar 1;36(2):91-98. doi: 10.1097/MCA.0000000000001459. Epub 2024 Nov 27. PMID 39601687

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total 51 subjects were enrolled in the CVT-ISR study at nine (9) investigational sites in Europe between October 20, 2021, and April 21, 2022.
Period: Overall Study
Arm/Group | Drug Eluting Balloon
Started | 51
Completed | 50
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Drug Eluting Balloon
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.2 (11.2)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 38
  Female | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 27
  More than one race | 0
  Unknown or Not Reported | 18
Prior Percutaneous coronary revascularization (Prior PCI) [Count of Participants; unit: Participants] | 51

OUTCOME MEASURES:

1. Primary Outcome: The Primary Safety Endpoint for the CVT-ISR Study: Freedom From Target Lesion Failure (TLF) Rate
Description: Composite rate of cardiovascular death, target vessel myocardial infarction and clinically-driven target lesion revascularization (TLR).
Time Frame: 6 months post-index procedure
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Drug Eluting Balloon
Number analyzed (Participants) | 51
Participants
  Target Lesion Failure | 4
  Cardiovascular Death | 1
  Target Vessel MI | 0
  Clinically-Driven Target Lesion Revascularization | 3

2. Primary Outcome: The Primary Effectiveness Endpoint for the CVT-ISR Study: In-stent Late Lumen Loss (LLL)
Description: In-Stent Late Lumen Loss (LLL) measures the reduction in the luminal diameter of a stented artery over a specified period after stent implantation, typically assessed using angiographic imaging. The unit of measurement for this outcome is expressed in millimeters (mm) or percentage (%), depending on the reporting method. The LLL is calculated by comparing the luminal diameter at a follow-up time point to the post-procedure luminal diameter.
Time Frame: 180 days post-procedure
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Drug Eluting Balloon
Number analyzed (Participants) | 51
millimeters (mm) | 0.40 (0.48)

3. Secondary Outcome: Composite Rate of Target Lesion Failure (TLF)
Description: TLF is defined as composite rate of cardiovascular death, target vessel myocardial infarction and clinically-driven target lesion revascularization (TLR).
Time Frame: 30 days post-procedure and 12 months
Population: Analysis population includes all intent to treat (ITT) patients with cardiovascular death, target vessel MI and clinically-driven TLR cumulative at each timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Drug Eluting Balloon
Number analyzed (Participants) | 51
Participants
  30 days post-procedure | 1
  12 months | 5

4. Secondary Outcome: Composite Rate of Target Vessel Failure (TVF)
Description: Target vessel failure (TVF) is defined as composite rate of cardiovascular death, target vessel myocardial infarction, and clinically-driven target vessel revascularization (TVR).
Time Frame: 30 days post-procedure, 180 days and 12 months
Population: Analysis population includes all intent to treat (ITT) patients with cardiovascular death, target vessel MI and clinically-driven TVR cumulative at each timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Drug Eluting Balloon
Number analyzed (Participants) | 51
Participants
  30 days post-procedure | 1
  180 days | 7
  12 months | 9

5. Secondary Outcome: Clinically Driven Target Lesion Revascularization (TLR)
Description: TLR is defined as any repeat PCI of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion.
Time Frame: 12 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Drug Eluting Balloon
Number analyzed (Participants) | 51
Participants | 4

6. Secondary Outcome: Clinically-driven Target Vessel Revascularization (TVR)
Description: TVR is defined as any repeat percutaneous intervention or surgical bypass of any segment of the target vessel including the target lesion.
Time Frame: 180 days and 12 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Drug Eluting Balloon
Number analyzed (Participants) | 51
Participants
  180 days | 5
  12 months | 7

7. Secondary Outcome: Rate of Vascular Access Site Complications
Description: The rate of vascular access site complications is defined as the combined rate of hematoma, AV fistula or a pseudoaneurysm that required intervention, such as surgical repair, transfusion or a prolonged hospital stay or requiring a new hospital admittance.
Time Frame: 12 months
Population: Analysis population includes all intent to treat (ITT) patients with access site complications of Hematoma, AV Fistula or Pseudoaneurysm.
Measure: Count of Participants; unit: Participants
Arm/Group | Drug Eluting Balloon
Number analyzed (Participants) | 51
Participants
  Hematoma | 0
  AV Fistula | 0
  Pseudoaneurysm | 0

8. Secondary Outcome: Lesion Success:
Description: Lesion success, defined as achievement of a final in-lesion residual diameter stenosis of <30% (by QCA), using any device after wire passage through the lesion.
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Drug Eluting Balloon
Number analyzed (Participants) | 51
Participants | 50

9. Secondary Outcome: Technical Success
Description: Technical success, defined as achievement of a final in-lesion residual diameter stenosis of <30% (by QCA), using the CVT Everolimus coated PTCA Catheter without a device malfunction after wire passage through the lesion.
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Drug Eluting Balloon
Number analyzed (Participants) | 51
Participants | 47

10. Secondary Outcome: Clinical Success (Per Subject)
Description: Clinical success (per subject) defined as technical success without the occurrence of major adverse cardiac events during the procedure.
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Drug Eluting Balloon
Number analyzed (Participants) | 51
Participants | 48

11. Secondary Outcome: Procedural Success
Description: Procedural success (per subject) defined as lesion success without the occurrence of major adverse cardiac events during the procedure.
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Drug Eluting Balloon
Number analyzed (Participants) | 51
Participants | 50

ADVERSE EVENTS:
Time Frame: 12 Months
Arm/Group | Drug Eluting Balloon
All-Cause Mortality (participants affected / at risk) | 1/51
Serious Adverse Events (participants affected / at risk) | 25/51
Other Adverse Events (participants affected / at risk) | 21/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Drug Eluting Balloon (N=51)
Restenosis, non-target lesion (Cardiac disorders) | 4
Angina, Unstable (Cardiac disorders) | 2
Stroke Suspicion (Cardiac disorders) | 1
Stable angina (Cardiac disorders) | 1
CABG, non-treated lesion (Cardiac disorders) | 1
CABG, target vessel (Cardiac disorders) | 1
Coronary Artery Restenosis (Injury, poisoning and procedural complications) | 5
Procedural Dissection (Injury, poisoning and procedural complications) | 1
Chest Pain (General disorders) | 1
Sternal wound (General disorders) | 1
Thoracic Pain (General disorders) | 1
Sudden Death, unknown cause (General disorders) | 1
Death, failure to thrive (General disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
GI Bleeding (Gastrointestinal disorders) | 1
Abdominal Aorta Aneurysm (Vascular disorders) | 1
Lower Limb Ischemia (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Drug Eluting Balloon (N=51)
Thoracic pain (General disorders) | 4
Chest pain (General disorders) | 3
Hypertension (General disorders) | 1
Non-cardiovascular death (General disorders) | 1
Positive stress test (General disorders) | 1
Post-surgical injury (General disorders) | 1
Sternal wound (General disorders) | 1
Angina, stable (Cardiac disorders) | 3
Restenosis, non-treated lesion (Cardiac disorders) | 3
Bradycardia (Cardiac disorders) | 1
Stroke suspicion (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Lower limb ischemia (General disorders) | 2
Temporary hand/leg paralysis (General disorders) | 1
Target lesion restenosis (General disorders) | 1
Coronary artery restenosis (Injury, poisoning and procedural complications) | 3
Procedural dissection (Injury, poisoning and procedural complications) | 1
Urinary tract infection (Renal and urinary disorders) | 1
Erectile dysfunction (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
GI bleeding (Gastrointestinal disorders) | 1
Skin/Rash infection (Infections and infestations) | 2
Covid 19 (Infections and infestations) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1
Cutaneous hemorrhage (Skin and subcutaneous tissue disorders) | 1
Erysipelas (Skin and subcutaneous tissue disorders) | 1
Diabetes (Metabolism and nutrition disorders) | 1
Faintness (Nervous system disorders) | 1
Gingivorrhagia (General disorders) | 1
Abdominal aorta aneurysm (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-22): https://cdn.clinicaltrials.gov/large-docs/00/NCT05731700/Prot_SAP_000.pdf